CLINICAL TRIAL: NCT01324297
Title: The Topical Niacin Skin Flush Test: A Means for Longitudinal Monitoring of Two Different Biological Subgroups of Patients With First Episode Psychosis
Brief Title: The Topical Niacin Skin Flush Test in First Episode Psychosis
Status: Terminated | Type: Observational
Why Stopped: Unable to secure funding for second phase of study (i.e., niacin skin flush test in early psychosis patients).
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Beverly Butler, Research Neuropsychologist, Nova Scotia Health Authority
Other Study IDs: CDHA-RS_2011-215
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Diagnostic Techniques and Procedures; Sensitivity and Specificity; Skin Tests; Biological Markers
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Control: Caucasian males and females between 19 and 30 years of age.
  Interventions: Other: skin test
- First Episode Psychosis: Caucasian males and females between 19 and 30 years of age within twelve months of initial DSM IV TR diagnosis of schizophreniform psychosis, schizophrenia, schizoaffective disorder or psychotic disorder NOS.
  Interventions: Other: skin test

INTERVENTIONS:
Other: skin test — four patches of 2 x 3cm thin blotting paper will be soaked with an equivalent amount (0.1 mL) of aqueous methyl nicotinate in four different concentrations: 0.1, 0.01, 0.001, 0.0001 M. The four patches will then be applied at the same time to the inner forearm for 60 seconds.

SUMMARY:
The purpose of this study is to gather normative data from healthy adults and to determine a sensitive and specific cut-off value for responders and non-responders to the Niacin Skin Flush Test in a sample of first episode psychosis patients.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* within twelve months of initial DSM IV TR diagnosis of schizophreniform psychosis, schizophrenia, schizoaffective disorder or psychotic disorder NOS
* outpatient

Exclusion Criteria:

* known allergy to study compound (methyl nicotinate, vitamin B3, niacin)
* skin conditions (e.g., dermatitis, psoriasis, eczema)
* diagnosis or treatment for medical conditions that may affect normal vascular tone (e.g., diabetes, vasculitis, chronic hypertension, etc.)
* Use of anti-inflammatory, antibiotic, or antihistamine medications within one month prior to study entry
* Use of supplements like Omega 3 fatty acids within 3 months prior to study entry
* Use of vitamin or nutritional supplement containing a dose of niacin/nicotinic acid above 50 mg/day at study entry

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2011-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in visual rating of skin response (redness and oedema) | ratings made at 3, 6, 9 and 12 minutes after application of methyl nicotinate
  A 7-point visual rating scale, previously tested for reliability (Kerr 2008), to visually rate the skin response to aqueous methyl nicotinate (niacin) with respect to both redness and oedema as a function of increasing niacin concentrations.Ratings will be acquired every three minutes over a 12-minute period starting at the time of solution application.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip G Tibbo, MD, FRCPC, Study Chair — Capital District Health Authority, Nova Scotia, Canada
Locations (1):
- Nova Scotia First Episode Psychosis Program; QEII health Sciences Centre; Capital District Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Kerr M, Cotton S, Proffitt T, McConchie M, Markulev C, Smesny S, McGorry P, Berger G. The topical niacin sensitivity test: an inter- and intra-rater reliability study in healthy controls. Prostaglandins Leukot Essent Fatty Acids. 2008 Jul-Aug;79(1-2):15-9. doi: 10.1016/j.plefa.2008.06.001. Epub 2008 Jul 24. PMID 18656334
- [Background] Nadalin S, Buretic-Tomljanovic A, Rubesa G, Tomljanovic D, Gudelj L. Niacin skin flush test: a research tool for studying schizophrenia. Psychiatr Danub. 2010 Mar;22(1):14-27. PMID 20305586